CLINICAL TRIAL: NCT00766376
Title: Safety and Efficacy Evaluation of Fractional Erbium Treatment
Brief Title: Safety and Efficacy Evaluation of Erbium Treatment
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Palomar Medical Technologies, Inc. (Industry)
Responsible Party: Medical Director, Palomar Medical Technologies, Inc.
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ERf-02
Record Dates: First submitted 2008-09-30; First posted 2008-10-03 (Estimated); Results first posted 2010-01-29 (Estimated); Last update posted 2010-01-29 (Estimated); Status verified 2010-01

CONDITIONS: Skin Aging
MeSH Terms: interventions — Lasers, Solid-State

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Erbium laser — Erbium laser treatment. Each subject will undergo up to 6 treatment sessions

SUMMARY:
The purpose of this research study is to evaluate the safety and effectiveness of erbium lasers for dermatological cosmetic procedures.

DETAILED DESCRIPTION:
The purpose of this investigation is to evaluate erbium laser devices for dermatological cosmetic procedures.

Each subject will undergo up to 6 treatment sessions, with scheduled time-points for follow-up visits. The Investigator determines the number of treatments. Subjects may be treated on there face, neck, chest or other body areas as deemed appropriate by the Investigator. At each visit, the treated areas will be clinically evaluated for side effects and will also have photographs taken of their treated areas. Subjects will be asked to complete a self-assessment questionnaire at different time points throughout their study participation.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female Adults (18 years or older).
* Subjects who can read, understand, and sign the Informed Consent Form.
* Subjects willing and able to comply with all study requirements.

Exclusion Criteria:

* Subjects with active localized or systemic infections.
* Immunocompromised subjects.
* Subjects with coagulation disorder.
* History of skin photo sensitivity disorders, or use of photosensitizing drugs (e.g., tetracycline or sulfa drugs).
* Pregnant and/or lactating (All female volunteers will be advised about using birth control during the period of study).
* In the opinion of the trained clinician, subject is unwilling or unable to adhere to all study requirements, including application and follow-up visits.
* Use of Accutane® within the past 6 months.
* Subjects with a history of radiation therapy to the treatment area.
* Subjects with any skin pathology or condition that could interfere with evaluation or with the use of typical ancillary medical treatments or care used before, during or after treatments.
* Subjects have undergone dermatological procedures (e.g., laser or light treatments) for the treatment of wrinkles, skin resurfacing, or skin rejuvenation in the treatment area within 1 year of study participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 151 (Actual)
Dates: Start 2007-07; Primary Completion 2009-07 (Estimated); Study Completion 2009-07 (Estimated)

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Scripps Clinic Laser & Cosmetic Dermatology, San Diego, California
  - Palomar Medical Technologies, Inc., Burlington, Massachusetts
  - Brooke Seckel, MD, Concord, Massachusetts
  - Skin & Laser Surgery Center, Nashua, New Hampshire
  - The University of Texas Southwestern Medical Center at Dallas, Dallas, Texas

RESULTS

PARTICIPANT FLOW:
Groups:
- Erbium Laser: Each Subject will undergo 1 - 6 treatment sessions, with 5 scheduled time-points for follow-up visits. Additional follow-up visits may be required to accommodate optional biopsies or to evaluate any concerns related to the course of healing. At each visit, the treated areas will be clinically evaluated and photographed.
Period: Overall Study
Arm/Group | Erbium Laser
Started | 151
Completed | 124
Not Completed | 27
Not completed — Withdrawal by Subject | 27

BASELINE CHARACTERISTICS:
Groups:
- Erbium Laser: Each subject will undergo a minimum of 1 treatment with 5 scheduled follow-up visits. Additional follow-up visits may be required to accommodate optional biopsies or to evaluate any concerns related to the course of healing. At each visit, the treated areas will be clinically evaluated and photographed.
Arm/Group | Erbium Laser
Number analyzed (Participants) | 124
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 113
  >=65 years | 11
Age Continuous [Mean (Standard Deviation); unit: years] | 55 (8.11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 116
  Male | 8
Region of Enrollment [Number; unit: participants]
  United States | 124

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants That Scored Above a One Category (Mild) Improvement Using the Fitzpatrick Wrinkle Scale.
Description: To assess wrinkle improvement, 3 blinded evaluators use the validated Fitzpatrick Wrinkle Scale (FWS), a 0 to 9 (0=no wrinkles, 9=severe wrinkles) point scale to score the degree of wrinkles, fine lines, and the severity of skin elastosis. Evaluators assign a FWS score to pre-treatment and post-treatment photographs. The difference between the two scores is the amount (i.e., category) of wrinkle improvement. An improvement of one category means a mild improvement in wrinkle reduction.
Time Frame: participants at three months
Measure: Number; unit: Participants
Arm/Group | Erbium Laser
Number analyzed (Participants) | 151
Participants | 124

2. Secondary Outcome: Number of Participants That Have Reduction in Pigmented Lesions and Dyschromia.
Description: To assess reductions in pigmented lesions and dyschromia, blinded evaluators were asked to assess pre-treatment and post-treatment photographs. The blinded evaluators were asked to grade percent improvement for pigmentation using a 0 to 10 scale (0=none and 10=severe) and the following quartile improvement scale: 1=1-24%, 2=25-49%, 3=50-74% and 4=75-100%. The blinded-evaluator scores were tabulated and analyzed in order to assess the effects.
Time Frame: participants at three months
Measure: Number; unit: Participants
Arm/Group | Erbium Laser
Number analyzed (Participants) | 151
Participants | 124

ADVERSE EVENTS:
Time Frame: Minimum of 3 months post treatment, or until adverse events resolve
Arm/Group | Erbium Laser
Serious Adverse Events (participants affected / at risk) | 0/124
Other Adverse Events (participants affected / at risk) | 124/124
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Erbium Laser (N=124)
Petechiae (Skin and subcutaneous tissue disorders) | 26 — Transient side effects all resolved.
Edema (Skin and subcutaneous tissue disorders) | 123 — Transient side effects all resolved.
Erythema (Skin and subcutaneous tissue disorders) | 124 — Transient side effects all resolved.
Bleeding (Skin and subcutaneous tissue disorders) | 98 — Transient side effects all resolved.
Oozing (Skin and subcutaneous tissue disorders) | 71 — Transient side effects all resolved.
Skin Texture Changes (Skin and subcutaneous tissue disorders) | 9 — Transient side effects all resolved.
Bronzing (Skin and subcutaneous tissue disorders) | 67 — Transient side effects all resolved.
Sloughing (Skin and subcutaneous tissue disorders) | 55 — Transient side effects all resolved.
Shrinkage (Skin and subcutaneous tissue disorders) | 9 — Transient side effects all resolved.
Increased Sensitivity (Skin and subcutaneous tissue disorders) | 40 — Transient side effects all resolved.
Crusting (Skin and subcutaneous tissue disorders) | 55 — Transient side effects all resolved.
Hyperpigmentation (Skin and subcutaneous tissue disorders) | 35 — Transient side effects all resolved.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No